CLINICAL TRIAL: NCT00033124
Title: Behavioral Trial for the Treatment of Methamphetamine Dependence
Brief Title: A Behavioral Trial for the Treatment of Methamphetamine Dependence. - 1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-CTO-0009-1; NCT00024739 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2003-08

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Behavior Therapy

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to examine behavioral treatment for methamphetamine dependence.

DETAILED DESCRIPTION:
To characterize meth. withdrawal symptoms using a multidimensional withdrawal questionnaire; to field test and investigate the effect of using an algorithm developed for discriminating between new use and residual carry-over of meth metabolites in urine and to evaluate the treatment response of meth. users to participation in the thrice weekly psychosocial protocol to be used as a "platform" in future pharmacotherapy trials.

ELIGIBILITY:
Inclusion Criteria:

Male or Female at least 18 yrs of age; DSM-4 diagnosis of methamphetamine (METH) dependence; be willing to comply with study procedures; verbalize understanding of consent and provide written consent and willingness to complete study procedures; be seeking treatment for METH dependence.

Exclusion Criteria:

Additional criteria available during screening at the site.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2001-07; Study Completion 2002-06

PRIMARY OUTCOMES:
Withdrawal symptoms
New Use algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rawson, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (5):
- United States (5):
  - South Bay Treatment Center, Chula Vista, California
  - Matrix Institute on Addictions, Costa Mesa, California
  - John A. Burns School of Medicine, Honolulu, Hawaii
  - Powell Chemical Dependency Center, Des Moines, Iowa
  - Comprehensive Mental Health Services, Inc, Independence, Missouri